CLINICAL TRIAL: NCT02019537
Title: Allogeneic Platelet-Rich Plasma Versus Corticosteroid Injection for the Treatment of Rotator Cuff Disease: A Randomized Controlled Trial
Brief Title: Subacromial Injection of Allogeneic Platelet Rich Plasma (PRP) for Shoulder Impingement Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hyunchul Jo, Associate Professor, SMG-SNU Boramae Medical Center, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BRM-13-01
Record Dates: First submitted 2013-12-18; First posted 2013-12-24 (Estimated); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Shoulder Impingement Syndrome
MeSH Terms: conditions — Shoulder Impingement Syndrome

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- Steroid group (Active Comparator): Triamcinolone injection group
  Interventions: Procedure: Steroid injection into the subacromial space
- PRP group (Experimental): Allogeneic PRP injection group
  Interventions: Procedure: Allogeneic PRP injection into the subacromial space

INTERVENTIONS:
Procedure: Steroid injection into the subacromial space — * Group: Steroid
  * Total volume of injection drugs: 4ml(1ml of triamcinolone acetonide 40mg/ml + 3ml of 2% lidocaine)
  * The number of injections : only once during the study period
  * Injection site : subacromial space
  * Material : 25-gauze spinal needle
  * Subacromial injections were performed using ultrasonographic guidance.
  Arms: Steroid group
Procedure: Allogeneic PRP injection into the subacromial space — * Group: Allogeneic PRP
  * Total volume of injection drugs: 4ml
  * The number of injections : only once during the study period
  * Injection site : subacromial space
  * Material : 25-gauze spinal needle
  * Subacromial injections were performed using ultrasonographic guidance.
  Arms: PRP group

SUMMARY:
The purpose of this study is to investigate the efficacy of allogeneic PRP in patients with subacromial impingement disease

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 years of age and older
* Patients who have unilateral shoulder pain.
* Patients who have had pain at least for 3 months
* To be included in the study- participants are required to have a & b.(mentioned below)

  1. Pain with one of the two tests

     * Neer's sign: passive overpressure at full shoulder flexion with the scapula fixed
     * Hawkins test: passive internal rotation at 90 degree of shoulder flexion in the scapular plane and in progressive degree of horizontal adduction
  2. Pain with one of the two tests

     * Painful arc: active shoulder abduction
     * Jobe's test: The examiner passively elevates the patient's shoulder to 90 degrees of abduction with internal rotation. The examiner then applies a downward pressure against the arm

Exclusion Criteria:

* Patients who received any drug by subacromial injection for treatment within 3 months prior to this enrollment.
* Patients who have a history of shoulder trauma including dislocation- subluxation- and fracture- breast cancer- or surgery around shoulder- neck and upper back
* Patients who have a isolated acromioclavicular joint pathology
* Patients who have a full-thickness rotator cuff tear (evidenced by MR or ultrasonography)
* Patients with symptomatic cervical spine disorders
* Patients who have a History of allergic adverse reactions to corticosteroid
* Patients are unable to give informed consent to participate in the study
* Patients are unable to come into the clinic for regular follow-up
* Patients with adhesive capsulitis- acromioclavicular arthropathy- polyarthritis- infectious arthritis- rheumatoid arthritis or diagnosed fibromyalgia
* Patients with concurrent bilateral shoulder pain
* Patients with neurological deficit
* Patients who have severely abnormal radiological findings including malignancy, severe osteoarthritis of the glenohumeral joint, severe skeletal abnormalities decreasing the subacromial space and etc.
* Presence of shoulder pain with limitation of both active and passive movements of the glenohumeral joint of 25% in at least 2 directions (abduction, flexion, external rotation, internal rotation), as compared with the contralateral shoulder or with normal values
* Patients with Diabetes mellitus
* Patients taking anticoagulants
* Pregnant women or lactating mothers
* Patients who are difficulty participating in data collection due to communication problem and serious mental illness
* Patients with serious condition which can affect this study such as severe cardiovascular diseases- renal diseases- liver diseases- endocrine diseases- and cancers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-02; Primary Completion 2016-06 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Safety determined with symptoms & signs of infection and immune response and adverse events evaluated with NCI-CTCAE v3.0 | Postinjection 1month
  Presence of general symptoms or signs associated with infection and immune response, such as rash, pruritus, fever, chills, urticaria, or dyspnea.
  Injection sites were examined to identify erythema, swelling, or abnormal discharge.
  Adverse events were categorised with use of the National Cancer Institute Common Terminology Criteria for Adverse Events scale, version 3.0.
Constant-Murley score | Postinjection 1month
  The Constant-Murley score (CMS) is a 100-points scale composed of parameters defining the level of pain and the ability of performing daily activities.

CONTACTS AND LOCATIONS:
Locations (1):
- Joint & Spine Center, SMG-SNU Boramae Medical Center, Department of Orthopedic Surgery, Seoul National University College of Medicine, Seoul, South Korea